CLINICAL TRIAL: NCT06829615
Title: Contactless Measurement of Heart Rate, Heart Rate Variability, Breathing Rate and Blood Pressure Using Face Video Analysis (Remote Photoplethysmography) - Validation of Shen.AI Software
Brief Title: Contactless Measurement of Heart Rate, Heart Rate Variability, Breathing Rate and Blood Pressure Using Remote Photoplethysmography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SHEN.AI spółka z ograniczoną odpowiedzialnością oddział w Polsce (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MDF-01-008-03
Record Dates: First submitted 2025-02-10; First posted 2025-02-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Heart Rate; Heart Rate Variability; Breathing Rate; Blood Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HR, HRV, BR, and BP measured using Shen.AI and reference methods (Experimental)
  Interventions: Device: Shen.AI

INTERVENTIONS:
Device: Shen.AI — Contactless measurement of heart rate, heart rate variability, breathing rate, and blood pressure using Shen.AI software and reference methods.

SUMMARY:
The purpose of this study it to evaluate the accuracy of heart rate, heart rate variability, breathing rate and blood pressure measurement with the use of Shen.AI software.

DETAILED DESCRIPTION:
The primary objective of this clinical study is to assess the accuracy of heart rate (HR), heart rate variability (HRV), breathing rate (BR), and blood pressure (BP) measurements obtained using Shen.AI software as the investigational device under its intended conditions of use, enabling users to obtain reliable information about their physiological state. These conditions include measurements taken at rest, in a home-like environment, with participants independently operating a mobile device or laptop equipped with a camera.

Physiological parameters, including HR, HRV, BR, and BP, will be measured and estimated using remote photoplethysmography (rPPG) based on a 1-minute facial video analysis processed by Shen.AI software.

Throughout all measurements, participants will be connected to a reference device that records ECG while simultaneously measuring chest impedance (impedance pneumography). Additionally, each participant will wear a respiratory belt transducer. Depending on the measurement type, the participant's blood pressure will be assessed using either an auscultatory or an automatic blood pressure monitor. The study will be conducted on a diverse group of participants, varying in blood pressure, gender, age, skin phototype, and BMI.

For each measured parameter, results obtained from both methods will be compared using Bland-Altman analysis or non-parametric limits of agreement.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to read and write in Polish or English
* Ability to operate a mobile device and a laptop without requiring glasses
* Ability to understand the study procedure
* Ability to communicate and follow instructions from the study personnel
* Provision of written informed consent for participation in the study and for the processing of personal data by the research team and the study sponsor
* Blood pressure values in accordance with the distribution of the study group

Exclusion Criteria:

* Pregnancy
* Age below 18 years
* Failure to provide the required information in the participant's informational questionnaire
* Non-compliance with the study procedure or instructions from the study personnel
* Extensive facial skin damage (e.g., abrasions, wounds, burns)
* A disease process affecting a significant portion of the face
* Extensive facial dressing
* Extensive facial tattoos or facial painting
* Significant facial deformity (e.g., tumor)
* Inability to maintain a stable head position during measurement
* Persistent cough preventing stillness during measurement
* Respiratory dysfunction such as dyspnea, irregular or shallow breathing
* Diagnosed arrhythmia (except for sinus bradycardia or sinus tachycardia)
* Moderate or severe anemia
* Diagnosed conditions such as left ventricular systolic dysfunction, aortic valve stenosis, or other cardiac or circulatory diseases leading to low stroke volume, low pulse amplitude, or pulsus paradoxus
* Implanted cardiac pacemaker
* Blood pressure difference between arms exceeding 15 mmHg for systolic pressure or 10 mmHg for diastolic pressure
* Inability to determine blood pressure in both arms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of the average heart rate (HR) measurement using the device under test compared to the reference measurement. | One appointment (day 1)
  Average HR will be estimated using Shen.AI software and compared with simultaneously recorded ECG .
Accuracy of the measurement of the heart rate variability index - Standard Deviation of Normal-to-Normal intervals (SDNN) using the device under test compared to the reference measurement. | One appointment (day 1)
  The heart rate variability index (SDNN) will be measured using Shen.AI software and compared with the simultaneously recorded ECG.
Accuracy of the breathing rate (BR) measurement using the device under test compared to the reference measurement. | One appointment (day 1)
  Average BR will be estimated using Shen.AI software and compared with the recorded impedance pneumography signal in the absence of read-out capability supported by the respiratory belt transducer.
Accuracy of systolic and diastolic blood pressure (BP) measurements using the device under test in relation to the reference measurement. | One appointment (day 1)
  Average BP will be estimated using Shen.AI software and compared with auscultatory blood pressure measurements.
Accuracy of systolic and diastolic blood pressure (BP) measurement using the device under test, taking into account the calibration of the BP measurement function, in relation to the reference measurement. | Two appointments (14 ± 3 days apart)
  Average BP will be estimated using Shen.AI software and compared with auscultatory blood pressure measurements. Measurements will be performed during two visits, with the second visit occurring 14 ± 3 days apart.

SECONDARY OUTCOMES:
Accuracy of the measurement of other heart rate variability metrics - Root Mean Square of Successive Differences (RMSSD) using the device under test. | One appointment (day 1)
  The heart rate variability index (RMSSD) will be measured using Shen.AI software and compared with the simultaneously recorded ECG.
Accuracy of blood oxygen saturation measurement using the device under test | One appointment (day 1)
  The blood oxygen saturation will be measured using Shen.AI software and compared with the simultaneously obtained blood oxygen measurements.
Accuracy of Body Mass Index (BMI) estimation using the device under test. | One appointment (day 1)
  The BMI will be measured using Shen.AI software and compared with the values obtained from a weight scale and stadiometer.

OTHER OUTCOMES:
Utility of the software under test for self-measurement of physiological parameters, as assessed by user and observer questionnaires. | One appointment (day 1)
  At the end of the appointment, two questionnaires will be used to assess the usability of the Shen.AI software.
  User Usability Questionnaire - completed by participants to evaluate the clarity of instructions, ease of use, calibration process, interface intuitiveness, perceived safety, and overall experience.
  Observer Usability Questionnaire - completed by study personnel to assess patient behavior, difficulties encountered during measurements, and potential usability issues.
  Each questionnaire consists of multiple-choice questions (e.g., "Very intuitive", "Intuitive", "Non-intuitive", "Very unintuitive") and open-ended questions. Higher-rated responses (e.g., "Very intuitive", "Intuitive") indicate better usability and user experience, while lower-rated responses suggest usability challenges or areas for improvement. Open-ended responses will be analyzed by a dedicated research team to identify key themes, usability issues, and potential improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Chojdak-Łukasiewicz, MD, PhD, Principal Investigator — Wroclaw Medical University
Locations (2):
- Poland (2):
  - OVO MEDICAL Sp. z o.o., Wroclaw, Lower Silesian Voivodeship
  - Przychodnia rehabilitacyjna R-MED, Wroclaw, Lower Silesian Voivodeship